CLINICAL TRIAL: NCT04450524
Title: Changing Eating Behavior Using Cognitive Training: A Randomized Clinical Trial
Brief Title: Changing Eating Behavior Using Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Comsa Loana, Principal Investigator, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phd Study 4
Record Dates: First submitted 2020-06-22; First posted 2020-06-29 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: Obesity; Overweight; Weight loss; Hypnosis; Food Inhibition Training; Go No Go Task
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will not know in which group they belong: intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnosis (Experimental): Hypnosis formed from hypnotic induction (an adapted version from Harvard Group Scale of Hypnotic Susceptibility) together with hypnotic suggestions about a future where they will control their eating behaviors by choosing the low-calorie food instead of dense calorie one.
  Interventions: Behavioral: Hypnosis
- Food Inhibition Training (Experimental): Participants will perform an online computer go-no-go task. They will be shown pictures of dense and low-calorie food together with neutral pictures, followed by the instruction to press or not a button when the pictures are framed in a bold frame (dense calorie food).
  Interventions: Behavioral: Food inhibition training
- Control (Placebo Comparator): Participants will perform an online computer go-no-go task. They will be shown pictures of dense and low-calorie food together with neutral pictures, followed by the instruction to press the button to indicate the position of the picture - left or right.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Hypnosis — Participants received hypnotic induction with hypnotic suggestions for their eating behaviors.
  Arms: Hypnosis
Behavioral: Food inhibition training — Training the associations between foods and motor inhibition using a GO-NO-GO computer task.
  Other Names: Food response inhibition training
  Arms: Food Inhibition Training
Behavioral: Control — A simple GO-NO-GO task
  Arms: Control

SUMMARY:
Obesity is a global health problem. New and more efficient interventions are needed to overcome this disease. This randomized clinical trial aims to evaluate the effectiveness of changing eating behavior using cognitive training. These types of interventions have the role of creating new routines (unconsciously processed), in terms of healthy eating behaviors.

DETAILED DESCRIPTION:
This is a randomized clinical trial with three groups. Participants will be found through social media announcements. The active interventions of cognitive training will be delivered at two groups: one group will receive through hypnosis and the other will receive through food inhibition training (a GO NO GO task). The control group will receive a simple GO NO GO task as an active placebo. The trial will be exclusively online and it consists of five sessions. Participants will complete their tasks on four Zoom sessions. Cognitive, emotional and behavioral data will be taken at four times: before the intervention starts, in the middle (after two sessions), at the end and at two follow up moments: one month and six months after the trial ends.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Persons who like high-calorie foods (self-report food preferences)
* Persons who have a medium to high score at the self-report daily snacking
* BMI>25

Exclusion Criteria:

* Enrolled in a weight loss program
* Under 18 years
* Health problems that can affect weight loss
* Persons with clinical problems such as diabetes, cardiovascular disease, mental problems, persons who take medicines that can affect weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline, pre-intervention; immediately after the intervention; 1 month; 6 month.
  Weight in kg
Change in Eating behaviour 1 - Daily Snacking | Baseline, pre-intervention; immediately after the intervention; 1 month; 6 month.
  A self reported questionnaire of high calorie food frequency
Change in Eating behaviour 2 - Quantity of calories intake | Baseline, pre-intervention; in the week of the intervention; 1 month; 6 month.
  A self reported diary of food in two different day of the week (weekday and weekend day)
Change in Eating behaviour 3 | Baseline, pre-intervention; immediately after the intervention;1 month; 6 month.
  Self-reported Three Factor Eating Questionnaire. The scale measures three aspects of eating behavior: cognitive restraint (CR), uncontrolled eating (UE), and emotional eating (EE). It has 21 items and the responses are on a four-point Likert scale ranging from 1 Definitely true to 4 Definitely false with three subscales one for each domain. Higher scores indicate greater CR, UE, or EE.

SECONDARY OUTCOMES:
Change in Positive and Negative Affect | Baseline, pre-intervention; during the intervention (after 2 days), immediately after the intervention;1 month; 6 month.
  Self-report - Positive and Negative Schedule (PANAS). The responses are made using Likert type ratings from 1 - Not at all, to 5 Very much. Higher scores on negative affect representing higher levels of negative affect and higher scores on positive affect representing higher levels of positive affect.
Change in Motivation | Baseline, pre-intervention; during the intervention (after 2 days), immediately after the intervention; 1 month; 6 month.
  Self-report - Intrinsic Motivation Inventory. The interest/enjoyment subscale is considered the self-report measure of intrinsic motivation; The responses are made using Likert type ratings from 1 - not at all true to 7 very true. Higher total scores indicate higher intrinsic motivation.
Change in Self-Efficacy | Baseline, pre-intervention; during the intervention (after 2 days), immediately after the intervention; 1 month; 6 month.
  Self-report - Weight Efficacy Lifestyle Questionnaire. The response is given using a Likert scale in 0 to10 points: 0 for "Not confident at all" and 10 indicates "Very confident". Higher total scores are associated with higher eating self-efficacy and motivation to make positive lifestyle changes.
Change in Eating Intentions | Baseline, pre-intervention; during the intervention (after 2 days), immediately after the intervention; 1 month; 6 month.
  Self-report - A three-point Likert scale created by authors. Higher scores indicate a stronger desire to eat high-calorie food.
Change in Eating Preferences | Baseline, pre-intervention; immediately after the intervention; 1 month; 6 month.
  Self-report - A three-point Likert scale created by authors about the preferences of high-calorie food. Higher scores mean a high preference for high-calorie food.

OTHER OUTCOMES:
Behavioral Activation | Baseline, pre-intervention.
  The Fun Seeking Subscale from the Behavioral Inhibition/Behavioral Activation Scales with 4 self-rated items using a 4-point Likert scale (1=very true for me, to 4=very false for me). Higher scores are linked to impulsivity.
Specific to food irrationality | Baseline, pre-intervention.
  Self report - Irrational Food Beliefs Scale. The responses are made using Likert type ratings from 1 - strongly disagree to 4 strongly agree. Highest scores are significantly associated with weight gain and poor weight loss maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Loana T Comsa, Phd Student, Principal Investigator — Babes-Bolyai University Cluj-Napoca
Locations (2):
- Romania (2):
  - Department of Clinical Psychology and Psychotherapy, Cluj-Napoca, Cluj
  - Departement of Clinical Psychology and and Psychotherapy, Babes-Bolyai University, Cluj-Napoca, Cluj

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams RC, Lawrence NS, Verbruggen F, Chambers CD. Training response inhibition to reduce food consumption: Mechanisms, stimulus specificity and appropriate training protocols. Appetite. 2017 Feb 1;109:11-23. doi: 10.1016/j.appet.2016.11.014. Epub 2016 Nov 9. PMID 27838443
- [Background] Haggard P, Cartledge P, Dafydd M, Oakley DA. Anomalous control: when 'free-will' is not conscious. Conscious Cogn. 2004 Sep;13(3):646-54. doi: 10.1016/j.concog.2004.06.001. PMID 15336254
- [Background] Haggard P. Human volition: towards a neuroscience of will. Nat Rev Neurosci. 2008 Dec;9(12):934-46. doi: 10.1038/nrn2497. PMID 19020512
- [Background] Houben K, Jansen A. Training inhibitory control. A recipe for resisting sweet temptations. Appetite. 2011 Apr;56(2):345-9. doi: 10.1016/j.appet.2010.12.017. Epub 2010 Dec 24. PMID 21185896
- [Background] Houben K, Jansen A. Chocolate equals stop. Chocolate-specific inhibition training reduces chocolate intake and go associations with chocolate. Appetite. 2015 Apr;87:318-23. doi: 10.1016/j.appet.2015.01.005. Epub 2015 Jan 13. PMID 25596041
- [Background] Jones A, Hardman CA, Lawrence N, Field M. Cognitive training as a potential treatment for overweight and obesity: A critical review of the evidence. Appetite. 2018 May 1;124:50-67. doi: 10.1016/j.appet.2017.05.032. Epub 2017 May 22. PMID 28546010
- [Background] Kirsch I, Lynn SJ. Hypnotic involuntariness and the automaticity of everyday life. Am J Clin Hypn. 1997 Jul;40(1):329-48. doi: 10.1080/00029157.1997.10403402. PMID 9265803
- [Background] Lawrence NS, O'Sullivan J, Parslow D, Javaid M, Adams RC, Chambers CD, Kos K, Verbruggen F. Training response inhibition to food is associated with weight loss and reduced energy intake. Appetite. 2015 Dec;95:17-28. doi: 10.1016/j.appet.2015.06.009. Epub 2015 Jun 29. PMID 26122756
- [Background] Oakley DA, Halligan PW. Hypnotic suggestion and cognitive neuroscience. Trends Cogn Sci. 2009 Jun;13(6):264-70. doi: 10.1016/j.tics.2009.03.004. Epub 2009 May 8. PMID 19428287
- [Background] Shallice T. Dual functions of consciousness. Psychol Rev. 1972 Sep;79(5):383-93. doi: 10.1037/h0033135. No abstract available. PMID 5076868
- [Background] Stice E, Lawrence NS, Kemps E, Veling H. Training motor responses to food: A novel treatment for obesity targeting implicit processes. Clin Psychol Rev. 2016 Nov;49:16-27. doi: 10.1016/j.cpr.2016.06.005. Epub 2016 Jul 21. PMID 27498406
- [Background] Strack F, Deutsch R. Reflective and impulsive determinants of social behavior. Pers Soc Psychol Rev. 2004;8(3):220-47. doi: 10.1207/s15327957pspr0803_1. PMID 15454347
- [Background] Turton R, Nazar BP, Burgess EE, Lawrence NS, Cardi V, Treasure J, Hirsch CR. To Go or Not to Go: A Proof of Concept Study Testing Food-Specific Inhibition Training for Women with Eating and Weight Disorders. Eur Eat Disord Rev. 2018 Jan;26(1):11-21. doi: 10.1002/erv.2566. Epub 2017 Nov 3. PMID 29098749
- [Background] Beck, I., Smits, D. J., Claes, L., Vandereycken, W., & Bijttebier, P. (2009). Psychometric evaluation of the behavioral inhibition/behavioral activation system scales and the sensitivity to punishment and sensitivity to reward questionnaire in a sample of eating disordered patients. Personality and Individual Differences, 47(5), 407-412
- [Background] Carver, C. S., & White, T. L. (1994). Behavioral inhibition, behavioral activation, and affective responses to impending reward and punishment: the BIS/BAS scales. Journal of personality and social psychology, 67(2), 319
- [Background] Giel KE, Speer E, Schag K, Leehr EJ, Zipfel S. Effects of a food-specific inhibition training in individuals with binge eating disorder-findings from a randomized controlled proof-of-concept study. Eat Weight Disord. 2017 Jun;22(2):345-351. doi: 10.1007/s40519-017-0371-3. Epub 2017 Mar 7. PMID 28271453
- [Background] Hofmann, W., Friese, M., & Wiers, R. W. (2008). Impulsive versus reflective influences on health behavior: A theoretical framework and empirical review. Health Psychology Review, 2(2), 111-137
- [Background] Norman, D. A., & Shallice, T. (1986). Attention to action. In Consciousness and self-regulation (pp. 1-18). Springer, Boston, MA.